CLINICAL TRIAL: NCT05834387
Title: The Impact of a Transitional Care Management Programme on the Migration Stress of Family Members of Patients Transferred Out of the EICU Under the "Health Care-family-environment" Linkage Model
Brief Title: The Impact of a Transitional Care Management Programme on the Migration Stress of Family Members of Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Xu Ren, Study Director, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Zunyi001
Record Dates: First submitted 2023-04-11; First posted 2023-04-28 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental)
  Interventions: Procedure: EICU Transfer Routine Care
- Experimental group (Experimental)
  Interventions: Procedure: Implementing interventions based on a 'health care-family-environment' linkage

INTERVENTIONS:
Procedure: EICU Transfer Routine Care — EICU Transfer Routine Care
  Arms: Control group
Procedure: Implementing interventions based on a 'health care-family-environment' linkage — Nursing interventions in the experimental group The interventions were based on the "health care-family-environment" linkage
  Arms: Experimental group

SUMMARY:
This study investigated the impact of the establishment and application of the "health care-family-environment" linkage mechanism on the level of migration stress, coping styles and care satisfaction of families of patients transferred from the EICU, in order to provide a reference for improving the physical and psychological health of families and to promote the role of family members in the social support of patients transferred out of this category.

ELIGIBILITY:
Inclusion Criteria:

1. Family members of trauma patients scheduled to be transferred from the EICU to a general unit within 24h;
2. Family members of patients aged ≥ 18 years;
3. Family members who are responsible for the main care tasks and medical decisions of the patient during hospitalisation;
4. Family members of patients with clear language and good communication skills;
5. Families of patients who volunteered to participate in this study.

Exclusion Criteria:

1. Family members of patients temporarily transferred out of the EICU or temporarily discharged from trauma
2. Families of patients who voluntarily request termination of treatment;
3. Family members of patients with cognitive impairment, speech impairment or mental abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Stress assessment | 48 hours
  Stress assessment assessed by ICU Transfer Stress Assessment Scale for Families of Patients Transferring Out

CONTACTS AND LOCATIONS:
Overall Officials: Xu Ren, Study Director — Zunyi Medical College
Locations (1):
- Zunyi Medical College, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No